CLINICAL TRIAL: NCT01101659
Title: A Double-Blind, 2-Way Crossover Study to Investigate the Effects of JNJ-40411813 on Ketamine-Induced Alterations in Neuropsychiatric Performance
Brief Title: Ketamine Challenge Study With JNJ-40411813
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CR017161
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Perceptual Disorders; Confusion; Schizophrenia
Keywords: Activity of JNJ-40411813; Challenge study
MeSH Terms: conditions — Perceptual Disorders; Confusion; Schizophrenia | interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone; Saline Solution; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): JNJ-40411813 500 mg as 20 mL of oral suspension single dose
  Interventions: Drug: JNJ-40411813
- 002 (Placebo Comparator): Placebo 20 mL of oral suspension single dose
  Interventions: Drug: Placebo
- 003 (Other): ketamine Ketanest S. vials of 20 ml with 5 mg/ml diluted with saline to 0.02 mg Ketamine per mL and per kg bodyweight of the volunteer
  Interventions: Drug: ketamine
- 004 (Other): normal saline infusion 0.5 mL /min over 90 minutes
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: JNJ-40411813 — 500 mg as 20 mL of oral suspension
  Arms: 001
Drug: normal saline — single dose
  Arms: 004
Drug: ketamine — 20 mL of oral suspension
  Arms: 003
Drug: Placebo — single dose
  Arms: 002

SUMMARY:
The objective of this study is to investigate whether JNJ-40411813 versus placebo reduces psychosis-like symptoms, induced by infusion of a low dose of ketamine. Effects of JNJ-40411813 on ketamine-induced symptoms will be evaluated about 3 hours after a single oral dose when the concentration of JNJ-40411813 in the blood is at its maximum and up to 24 hours after dose administration to assess the duration of a potential JNJ-40411813 effect.

DETAILED DESCRIPTION:
This will be a double-blind (neither physician nor the volunteer knowns whether placebo or active drug is administered), placebo-controlled, randomized (study drug is assigned by chance), 2-way crossover (the same procedure is repeated twice so that the volunteer receives placebo as well as active drug) study in cohorts of a maximum of 16 healthy male volunteers each, to investigate the effect of JNJ 40411813 or placebo on ketamine-induced psychosis-like symptoms. In the first cohort (Cohort 1), JNJ 40411813 effects at a dose level of 500 mg will be evaluated at the time of maximal plasma concentrations. If JNJ 40411813 significantly reduces psychotic symptoms relative to placebo, a second cohort (Cohort 2) will be initiated to investigate the effects of JNJ 40411813 at 24 hours following dose administration. If Cohort 1 shows no relevant effects of JNJ 40411813 the study will be stopped. If there are no relevant effects of JNJ 40411813 on the psychotic symptoms at 24 hours after dosing, a third cohort (Cohort 3) will be initiated to investigate the effects at 12 hours after dosing. If there are relevant effects of JNJ 40411813 at 24 hours after dosing, a fourth cohort (Cohort 4) following the same procedures as Cohort 1, will be initiated to investigate the effects at peak plasma concentration using a lower dose of JNJ 40411813. Volunteers will be randomly assigned in a crossover procedure to one of two sequences (JNJ 40411813/placebo or placebo/ JNJ 40411813) on Day -1 of the first study period of each cohort. At peak plasma level (Cohorts 1 and 4), 24 hours (Cohort 2) or 12 hours (Cohort 3) after dosing volunteers will receive ketamine as an infusion (i.e. directly into the vein) over 60 minutes. The ketamine administration will be preceded by a saline infusion over 90 minutes. Tests on the psychological function of the volunteers will be performed during and after saline and ketamine infusion. Safety assessments include daily ECG and vital signs, clinical laboratory assessments at the start and end of each study period, pulse oximetry (measurement of the oxygen content of the blood ) during each ketamine infusion and continuous Adverse Event Reporting. The study will be double blind for oral JNJ-40411813 or placebo, but open label (everyone knows the identity) for the IV administration of saline and ketamine. JNJ-40411813: 500 mg single oral dose or lower or matching placebo. Ketamine: continuous intravenous infusion of 0.005 mg/kg/min over 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2
* Nonsmokers
* Healthy on the basis of a psychiatric examination according to the MINI screen
* Healthy on the basis of clinical laboratory tests performed at screening
* Healthy on the basis of physical examination, vital signs (including standing blood pressure and heart rate) or 12 lead ECG at Screening

Exclusion Criteria:

* Having a contra-indication for the use of ketamine
* Significant history of or current psychiatric or neurological illness
* Positive urine screen for drugs of abuse at Screening or admission
* Positive alcohol breath test at Screening or admission
* History of alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of JNJ- 40411813 on ketamine-induced positive psychotic symptoms based on 4 items of the brief psychiatric rating scale (BPRS) in healthy male volunteers | 15 minutes after start of bolus injection of ketamine

SECONDARY OUTCOMES:
Investigate the effects of JNJ 40411813 on ketamine-induced negative symptoms,based on 3 items of the BPRS, dissociative effects (based on the 5-dimensions altered state of consciousness (5D-ASC), and cognitive performance | 15 min, 30 to 60 min after start of bolus injection of ketamine and at the end of ketamine infusion
Investigate the duration of action and the concentration-effect relationship of JNJ 40411813 | 3, 12 and 24 hours after dosing of JNJ 40411813
Investigate the safety, tolerability, and pharmacokinetics of JNJ 40411813 in healthy volunteers | During each Period on Days 1, 2 and 3 (if applicable) and at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Neuss, Germany

REFERENCES:
- [Derived] Salih H, Anghelescu I, Kezic I, Sinha V, Hoeben E, Van Nueten L, De Smedt H, De Boer P. Pharmacokinetic and pharmacodynamic characterisation of JNJ-40411813, a positive allosteric modulator of mGluR2, in two randomised, double-blind phase-I studies. J Psychopharmacol. 2015 Apr;29(4):414-25. doi: 10.1177/0269881115573403. Epub 2015 Mar 3. PMID 25735992
- [Derived] Kleinloog D, Uit den Boogaard A, Dahan A, Mooren R, Klaassen E, Stevens J, Freijer J, van Gerven J. Optimizing the glutamatergic challenge model for psychosis, using S+ -ketamine to induce psychomimetic symptoms in healthy volunteers. J Psychopharmacol. 2015 Apr;29(4):401-13. doi: 10.1177/0269881115570082. Epub 2015 Feb 17. PMID 25693889